CLINICAL TRIAL: NCT04061876
Title: Ruxolitinib in Combination With Corticosteroid as First Line Therapy for the Treatment of High Risk Acute Graft-Versus-Host Disease
Brief Title: First Line Therapy for High Risk Acute GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: LU DAOPEI MEDICAL (Unknown); 960th Hospital of PLA (Unknown); The Second Hospital of Hebei Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2019-177-01
Record Dates: First submitted 2019-08-17; First posted 2019-08-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: aGVHD; Stem Cell Transplant Complications
Keywords: aGVHD
MeSH Terms: interventions — ruxolitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ruxolitinib combined with Corticosteroids (Experimental): Participants began oral administration of ruxolitinib at 5 mg QD; Methylprednisolone: 1mg/kg/d , iv or iv gtt for at leas 5 days, then taper according to the clinical response.
  Interventions: Drug: Ruxolitinib; Drug: Corticosteroid
- Corticosteroids (Active Comparator): Methylprednisolone: 2mg/kg/d , iv or iv gtt for at least 1 week, then taper according to the clinical response.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Ruxolitinib — Participants began oral administration of ruxolitinib at 5 mg QD;Methylprednisolone: 1mg/kg/d , iv or iv gtt for at least 5 days, then taper according to the clinical response.
  Other Names: New
  Arms: Ruxolitinib combined with Corticosteroids
Drug: Corticosteroid — Methylprednisolone: 2mg/kg/d , iv or iv gtt for at least 3 days, then taper according to the clinical response. 1mg/kg/d , iv or iv gtt for at least 5 days, then taper according to the clinical response.
  Other Names: Traditional

SUMMARY:
The purpose of this study is to determine the efficacy and safety of combined Ruxolitinib With Corticosteroids as First Line Therapy for the Treatment of High risk aGVHD(acute graft-versus-host disease )

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGVHD) is treated with systemic corticosteroid immunosuppression as first line therapy. Many patients with high risk aGVHD do not respond to primary therapy, high-dose systemic corticosteroids; therefore, survival for those patients remains particularly poor. Here we determine the efficacy and safety of combined Ruxolitinib With Corticosteroids as First Line Therapy for the Treatment of High risk aGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with hematological diseases.
2. Have undergone first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies.
3. new onset of grade II~IV aGVHD or intermediate or high risk aGVHD (based on ST2, REG3a, other experimental objects) within 100 days post-transplantation.

Exclusion Criteria:

1. recipients of second allogeneic stem cell transplant.
2. acute GVHD induced by donor lymphocyte infusion, interferon.
3. received first line aGVHD treatment before enrollment.
4. overlap GVHD syndrome.
5. pregnant or breast-feeding women.
6. absolute neutrophil count (ANC) <0.5×10e9/L or platelet count (PLT) < 20×10e9/L
7. Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min measured or calculated by Cockroft-Gault equation.
8. uncontrolled infection
9. human immunodeficiency virus infection
10. active hepatitis b virus, hepatitis C virus infection and need antivirus treatment.
11. Subjects with evidence of relapsed primary disease, or subjects who have been treated for relapse after the allo-HSCT was performed, or graft rejection.
12. allergic history to Janus kinase inhibitors.
13. Severe organ dysfunction unrelated to underlying GVHD, including:

    Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction).

    Clinically significant or uncontrolled cardiac disease including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy.

    Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
14. Received Janus kinase inhibitor therapy after allo-HSCT for any indication.
15. Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) at Day 28 | Day 28 after treatment
  Defined as the proportion of participants demonstrating a complete response (CR), or partial response (PR).

SECONDARY OUTCOMES:
Six-month duration of response | Six-month after treatment
  Defined as the time from first response until graft-versus-host disease (GVHD) progression or death. Six-month duration of response will be assessed when all participants who are still on study complete the Day 180 visit.
Duration of response | Day 90 after treatment
  Defined as the time from first response until GVHD progression or death, when all participants who are still on study complete the Day 90 visit.
Nonrelapse mortality (NRM) | 2 years after treatment
  NRM was deﬁned as death from any cause without relapse. Cumulative incidence of NRM was analyzed in a competing risk framework using Gray's method.
Relapse rate | 2 years after treatment
  Defined as the proportion of participants whose underlying malignancy relapsed.Relapse was defined as hematologic recurrence of malignancies after transplantation. Cumulative incidence of relapse was analyzed in a competing risk framework using Gray's method.
Disease-free survival (DFS) | 2 years after treatment
  Defined as the time from first dose of ruxolitinib to the earliest date that a participant died, had a relapse/progression of the underlying malignancy, required additional therapy for aGVHD, or demonstrated signs or symptoms of chronic graft-versus-host disease (cGVHD).DFS will be evaluated in an intent-to-treat analysis by Kaplan Meier estimate and Log Rank test. Survival will be calculated from the date of randomization.
Overall survival (OS) | 2 years after treatment
  Defined as the time from study enrollment (first day of ruxolitinib treatment) to death due to any cause. OS will be evaluated in an intent-to-treat analysis by Kaplan Meier estimate and Log Rank test. Survival will be calculated from the date of randomization.
GVHD-free and relapse-free survival (GRFS) | 2 years after treatment
  GRFS was defined as the time onset of grade 3 to 4 aGVHD, moderate to severe cGVHD, or relapse/disease progression/death. GRFS will be evaluated in an intent-to-treat analysis by Kaplan Meier estimate and Log Rank test. Survival will be calculated from the date of randomization.
recurrence of aGVHD | 1 years after treatment
  Defined as the proportion of participants whose aGVHD relapsed.Relapse was defined as recurrence of new GVHD related symptoms after complete remission of aGVHD. Cumulative incidence of recurrence of aGVHD was analyzed in a competing risk framework using Gray's method.
Failure-free survival | 2 years after treatment
  Failure-free survival (FFS) refers to the time from randomization to disease relapse or progression, non-relapse mortality, or the addition of new therapy for aGVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Study Director — Chines PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuzmina Z, Eder S, Bohm A, Pernicka E, Vormittag L, Kalhs P, Petkov V, Stary G, Nepp J, Knobler R, Just U, Krenn K, Worel N, Greinix HT. Significantly worse survival of patients with NIH-defined chronic graft-versus-host disease and thrombocytopenia or progressive onset type: results of a prospective study. Leukemia. 2012 Apr;26(4):746-56. doi: 10.1038/leu.2011.257. Epub 2011 Sep 16. PMID 21926960
- [Background] Thepot S, Zhou J, Perrot A, Robin M, Xhaard A, de Latour RP, Ades L, Ribaud P, Petropoulou AD, Porcher R, Socie G. The graft-versus-leukemia effect is mainly restricted to NIH-defined chronic graft-versus-host disease after reduced intensity conditioning before allogeneic stem cell transplantation. Leukemia. 2010 Nov;24(11):1852-8. doi: 10.1038/leu.2010.187. Epub 2010 Sep 9. PMID 20827288
- [Background] Levine JE, Braun TM, Harris AC, Holler E, Taylor A, Miller H, Magenau J, Weisdorf DJ, Ho VT, Bolanos-Meade J, Alousi AM, Ferrara JL; Blood and Marrow Transplant Clinical Trials Network. A prognostic score for acute graft-versus-host disease based on biomarkers: a multicentre study. Lancet Haematol. 2015 Jan;2(1):e21-9. doi: 10.1016/S2352-3026(14)00035-0. Epub 2014 Dec 23. PMID 26687425
- [Background] Major-Monfried H, Renteria AS, Pawarode A, Reddy P, Ayuk F, Holler E, Efebera YA, Hogan WJ, Wolfl M, Qayed M, Hexner EO, Wudhikarn K, Ordemann R, Young R, Shah J, Hartwell MJ, Chaudhry MS, Aziz M, Etra A, Yanik GA, Kroger N, Weber D, Chen YB, Nakamura R, Rosler W, Kitko CL, Harris AC, Pulsipher M, Reshef R, Kowalyk S, Morales G, Torres I, Ozbek U, Ferrara JLM, Levine JE. MAGIC biomarkers predict long-term outcomes for steroid-resistant acute GVHD. Blood. 2018 Jun 21;131(25):2846-2855. doi: 10.1182/blood-2018-01-822957. Epub 2018 Mar 15. PMID 29545329
- [Background] von Bubnoff N, Ihorst G, Grishina O, Rothling N, Bertz H, Duyster J, Finke J, Zeiser R. Ruxolitinib in GvHD (RIG) study: a multicenter, randomized phase 2 trial to determine the response rate of Ruxolitinib and best available treatment (BAT) versus BAT in steroid-refractory acute graft-versus-host disease (aGvHD) (NCT02396628). BMC Cancer. 2018 Nov 19;18(1):1132. doi: 10.1186/s12885-018-5045-7. PMID 30453910
- [Derived] Dou L, Zhao Y, Yang J, Deng L, Wang N, Zhang X, Liu Q, Yang Y, Wei Z, Wang F, Jiao Y, Li F, Luan S, Hu L, Gao S, Liu C, Liu X, Yan J, Zhang X, Zhou F, Lu P, Liu D. Ruxolitinib plus steroids for acute graft versus host disease: a multicenter, randomized, phase 3 trial. Signal Transduct Target Ther. 2024 Oct 23;9(1):288. doi: 10.1038/s41392-024-01987-x. PMID 39438467
- [Derived] Dou L, Peng B, Li X, Wang L, Jia M, Xu L, Li F, Liu D. Ruxolitinib-corticosteroid as first-line therapy for newly diagnosed high-risk acute graft versus host disease: study protocol for a multicenter, randomized, phase II controlled trial. Trials. 2022 Jun 6;23(1):470. doi: 10.1186/s13063-022-06426-2. PMID 35668528
- [Derived] Yang JJ, Peng B, Fang S, Wei Y, Wang H, Zhao YX, Qian K, Wen YN, Liu DH, Dou LP. [Kinetics of MDSC in Patients Treated Steroids-Ruxolitinib as the First Line Therapy for aGVHD]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2022 Feb;30(1):276-285. doi: 10.19746/j.cnki.issn.1009-2137.2022.01.046. Chinese. PMID 35123640